CLINICAL TRIAL: NCT00838045
Title: A Prospective, Multi-Center Clinical Investigation to Evaluate the Safety & Effectiveness of the Bausch & Lomb AKREOS® TL (Model MI60) Intraocular Lens
Brief Title: Evaluation of the Safety & Effectiveness of the Bausch & Lomb AKREOS® TL Intraocular Lens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 451
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Cataract; Aphakia
MeSH Terms: conditions — Cataract; Aphakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Akreos TL intraocular lens (Experimental): Bausch & Lomb Akreos TL intraocular lens
  Interventions: Device: The Bausch & Lomb Akreos TL IOL (MI60) posterior chamber IOL

INTERVENTIONS:
Device: The Bausch & Lomb Akreos TL IOL (MI60) posterior chamber IOL — Surgery to implant the Bausch & Lomb Akreos TL Intraocular Lens will be performed using standard microsurgical techniques following cataract surgery.

SUMMARY:
This study is to evaluate the safety and effectiveness of the Bausch & Lomb Akreos TL (thin lens) intraocular lens (IOL) following implantation in adults requiring cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinically documented diagnosis of age-related cataract that is considered amenable to treatment with standard phacoemulsification/extracapsular cataract extraction.
* Subjects must be undergoing primary intraocular lens implantation for the correction of aphakia following continuous curvilinear anterior capsulotomy and phacoemulsification cataract extraction.
* Subjects must require a lens power from 15 to 30 diopters.
* Subjects must have a visual potential of 20/40 or better in the study eye.

Exclusion Criteria:

* Subjects with any anterior segment pathology for which extracapsular phacoemulsification cataract surgery would be contraindicated.
* Subjects with any inflammation or edema (swelling) of the cornea.
* Subjects with uncontrolled glaucoma or glaucoma under current treatment in the study eye or with ocular hypertension.
* Subjects with previous retinal detachment.
* Subjects with diabetic retinopathy (proliferative or non-proliferative).
* Subjects with rubella, bilateral congenital, traumatic, or complicated cataract.
* Subjects who have had previous ocular surgery in the planned operative eye, excluding ocular adnexa surgery.
* Subjects who have already received an Akreos TL IOL in the fellow eye.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Bast Corrected Visual Acuity | 24 months
  best-corrected visual acuity (BCVA)

SECONDARY OUTCOMES:
Uncorrected Visual Acuity | 24 months
Manifest Refraction | 24 Months
  mean manifest refraction

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kohnen, Principal Investigator — Klinikum der J.W. Goethe-Universität
Locations (1):
- Klinikum der J.W. Goethe-Universität, Frankfurt, Germany